CLINICAL TRIAL: NCT06487429
Title: Prospective, Phase II Clinical Study of Short Course Radiotherapy With Sequential Disitamab Vedotin Combined With S-1 and Sintilimab as Whole Course Neoadjuvant Therapy for HER2 Expressed Locally Progressive Gastric Cancer
Brief Title: Short Course Radiotherapy With Sequential Disitamab Vedotin Combined With S-1 and Sintilimab as Whole Course Neoadjuvant Therapy for HER2 Expressed Locally Progressive Gastric Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RCVDGIIIR015
Record Dates: First submitted 2024-06-27; First posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-05

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — S 1 (combination)

STUDY DESIGN:
Intervention Model Description: Single arm
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Short term radiotherapy with continuous use of Disitamab Vedotin, Sintilimab, and S-1 (Experimental): Short range radiotherapy, PCTV (Clinical Plan Target Area) DT 25Gy/5F, once daily for a total of 5 days, continuous irradiation, and IMRT (Intensity Modulated Radiotherapy) technology; After a week of rest, radiotherapy and chemotherapy combined with immunotherapy will be performed
  * Disitamab Vedotin: 2.5 mg/kg, intravenous infusion, d1，Q3W；
  * Sintilimab: 200mg, iv；
  * S-1: 40 mg/dose, oral, bid，d1-14；Q3W
  Interventions: Drug: Short range radiotherapy with sequential Disitamab Vedotin combined with S-1 and xindilizumab

INTERVENTIONS:
Drug: Short range radiotherapy with sequential Disitamab Vedotin combined with S-1 and xindilizumab — Short range radiotherapy, PCTV (clinical planned target area) DT 25Gy/5F, once a day, for a total of 5 days, continuous irradiation, and IMRT (intensity modulated radiation therapy) technology; After a week of rest, radiotherapy and chemotherapy combined with immunotherapy will be performed
  * Disitamab Vedotin: 2.5 mg/kg, intravenous infusion, d1, Q3W;
  * Sintilimab: 200mg, iv;
  * S-1: 40 mg/dose, oral, bid, d1-14; Q3W Whether to undergo adjuvant therapy after surgery is determined by the researcher

SUMMARY:
This study is a prospective, open label, phase II clinical study intended to include patients with locally advanced gastric adenocarcinoma who have not undergone any treatment and are eligible for surgery. The study aims to evaluate the efficacy and safety of the short course sequential radiotherapy regimen of Disitamab Vedotin combined with S-1 and Sintilimab in neoadjuvant therapy for HER2 expressing locally advanced gastric cancer.

DETAILED DESCRIPTION:
This study is a prospective, open label, phase II clinical study intended to include patients with locally advanced gastric adenocarcinoma who have not undergone any treatment and are eligible for surgery. The study aims to evaluate the efficacy and safety of the short course sequential radiotherapy regimen of Disitamab Vedotin combined with S-1 and Sintilimab in neoadjuvant therapy for HER2 expressing locally advanced gastric cancer.

After signing informed consent and screening to meet the inclusion criteria, the patient received full course neoadjuvant therapy: short course radiotherapy, rest for 1 week, sequential 3 cycles of Disitamab Vedotin combined with S-1 and Sintilimab, and preoperative imaging examination within 3-4 weeks after the last medication to evaluate the efficacy of neoadjuvant therapy and the possibility of curative D2 resection. The decision to undergo adjuvant treatment after radical surgery for gastric cancer is made by the researcher.

ELIGIBILITY:
Inclusion Criteria:

* 1. The subjects voluntarily joined this study, were able to complete the signing of the informed consent form, and had good compliance; 2. Age range from 18 to 75 years old (when signing the informed consent form), regardless of gender; 3. Gastric cancer or gastroesophageal junction adenocarcinoma confirmed by histology and/or cytology, diagnosed with local progression according to AJCC 8th edition standards, cT3-4N+M0 diagnosed with cTNM based on endoscopic ultrasound or enhanced CT/MRI scanning (combined with diagnostic laparoscopic exploration if necessary), and agreeing to undergo radical surgical treatment. The researcher evaluates the lesion as resectable; 4. Have not received systematic treatment for the current disease in the past, including anti-tumor radiotherapy, chemotherapy, immunotherapy, etc; 5. IHC results confirm HER2 expression (defined as IHC1+, 2+, 3+); 6. ECOG score 0-1 points; 7. Expected survival time ≥ 6 months; 8. The main organs are functioning well; 9. Fertility subjects must use appropriate methods of contraception during the study period and within 120 days after the end of the study. They must have a negative serum pregnancy test within 7 days before enrollment and must be non lactating subjects.

Exclusion Criteria:

-1. Diagnosed as malignant diseases other than gastric cancer within 5 years prior to initial administration (excluding curative basal cell carcinoma, squamous cell carcinoma of the skin, and/or curative resection of carcinoma in situ) 2. The tumor lesion has a tendency for bleeding (such as the presence of active ulcer tumor lesions with positive fecal occult blood test, history of vomiting blood or black stools within 2 months before signing the informed consent form, and a risk of gastrointestinal bleeding determined by the researcher), or having received blood transfusion treatment 4 weeks before the study medication; 3. Unable to take medication orally; 4. Currently participating in intervention clinical research treatment, or having received other research drugs or used research instruments within 4 weeks before the first administration; 5. Previously received the following therapies: anti-HER2, anti-PD-1, anti-PD-L1 drugs, anti-PD-L2 drugs, or drugs targeting another stimulus or synergistic inhibition of T cell receptors (including but not limited to CTLA-4, OX-40, CD137, etc.); 6. Have received systematic systemic treatment with traditional Chinese patent medicines and simple preparations with anti-tumor indications or drugs with immunomodulatory effect (including thymosin, interferon, interleukin, except for local use to control pleural effusion) within 2 weeks before the first administration; 7. Active autoimmune diseases that require systemic treatment (such as the use of disease relieving drugs, glucocorticoids, or immunosuppressants) have occurred within 2 years prior to the first administration. Alternative therapies (such as thyroid hormone, insulin, or physiological glucocorticoids used for adrenal or pituitary insufficiency) are not considered systemic treatments; 8. The study is currently undergoing systemic glucocorticoid therapy (excluding local glucocorticoids through nasal spray, inhalation, or other routes) or any other form of immunosuppressive therapy within 7 days prior to the first administration; Note: Physiological doses of glucocorticoids (≤ 10 mg/day of prednisone or equivalent) are allowed to be used; 9. Known allogeneic organ transplantation (excluding corneal transplantation) or allogeneic hematopoietic stem cell transplantation; 10. Known individuals who are allergic to the drugs used in this study; 11. Peripheral neuropathy ≥ grade 2; 12. Known history of human immunodeficiency virus (HIV) infection (i.e. HIV 1/2 antibody positive); 13. Active hepatitis B or hepatitis C subjects (HBsAg positive with HBV DNA titers higher than the upper limit of normal; HCVAb positive with HCV RNA titers higher than the upper limit of normal); 14. Have received a live vaccine within 30 days before the first administration (1st cycle, 1st day); Note: It is allowed to receive inactivated viral vaccines for seasonal influenza within 30 days before the first administration; However, it is not allowed to receive attenuated live influenza vaccines administered intranasally.

15. Pregnant or lactating women; 16. Existence of any serious or uncontrollable systemic diseases 17. Medical history or evidence of illness that may interfere with the trial results, hinder the full participation of subjects in the study, abnormal treatment or laboratory test values, or other situations that the researcher deems unsuitable for enrollment. The researcher believes that there are other potential risks that are not suitable for participation in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-05-08 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
pathological complete response (pCR) rate | an expected average of 4 months
  Pathological complete response rate (PCR) assessed by the blind independent Review Committee, defined as theabsence of viable tumour cells in the resected primary tumour specimen and all sampled regional lymph nodes(yPTONO)

SECONDARY OUTCOMES:
Overall Survival | an expected average of 5 years
  The time from the date of randomization to the death caused by any cause
RO resection rate | an expected average of 5mouths
  The rate of negative margin microscopically
dverse events (AEs) | an expected average of 5 years
  Adverse events and surgical safety
Primary pathological response (MPR) rate | an expected average of 1 years
  ≤ 10% residual live tumor
Disease free survival (DFS) | an expected average of 5 years
  The time from surgical resection to local recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Tao Zhang, MD, Principal Investigator — Union Hospital affiliated to Tongji Medical College of Huazhong University ofScience and Technology
Locations (1):
- Zhang Tao, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No